CLINICAL TRIAL: NCT01711983
Title: GORE® Septal Occluder Clinical Study: A Study to Evaluate Safety and Efficacy in the Treatment of Transcatheter Closure of Ostium Secundum Atrial Septal Defects (ASDs)
Brief Title: Safety and Efficacy of the GORE® Septal Occluder to Treat Ostium Secundum Atrial Septal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSO 10-09
Record Dates: First submitted 2012-10-11; First posted 2012-10-23 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Septal Defect, Atrial
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test Device (Experimental): ASD closure with the GORE® CARDIOFORM Septal Occluder
  Interventions: Device: GORE® CARDIOFORM Septal Occluder

INTERVENTIONS:
Device: GORE® CARDIOFORM Septal Occluder — Percutaneous Atrial Septal Defect Closure

SUMMARY:
The primary objective of the GORE® Septal Occluder Study is to evaluate the safety and efficacy of the occluder device in the treatment of transcatheter closure of ostium secundum atrial septal defects (ASDs). The data obtained in this study will evaluate this next generation device as compared to outcomes of prior studies conducted with the GORE® HELEX® Septal Occluder.

DETAILED DESCRIPTION:
Ostium secundum atrial septal defects present as a persistent communication between the atria and are a common congenital cardiac anomaly accounting for approximately 10% of all congenital heart disease. They are one of the most common congenital heart defects to present in adulthood. Untreated, ASDs produce right heart volume overload and progressive impairment over time, including reduced aerobic capacity, atrial dysrhythmias, congestive heart failure, pulmonary hypertension, and potential paradoxical embolism. In the U.S. alone it is estimated that approximately 10,000 new patients per year can be expected to have an ASD. Successful surgical repair of ASD has been performed for 50 years with continued improvement in technique and outcomes. King and Mills reported the first transcatheter closure of ASD in 1976, but the delivery system was quite large and impractical, especially for younger patients. With time, improvements in design concepts and materials discoveries have led to improved results in transcatheter closure systems. Several devices are now available commercially for transcatheter ASD closure.

ELIGIBILITY:
Inclusion Criteria:

* ASD less than or equal to 17 mm.

Exclusion Criteria:

* Conditions that would confound treatment of ASD or complicate distinguishing onset of adverse events.
* Unable to accommodate device delivery catheter.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Scott Lim, MD, Principal Investigator — University of Virginia, Children's Hospital Heart Center
Locations (1):
- University of Virginia, Children's Hospital Heart Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Device: ASD closure with the GORE® CARDIOFORM Septal Occluder
  Percutaneous Atrial Septal Defect Closure
Period: 6-Month Clinical Success Evaluation
Arm/Group | Test Device
Started | 400
Completed | 368
Not Completed | 32
Not completed — Missed Echocardiograph | 32
Period: 6-Month Closure Evaluation
Arm/Group | Test Device
Started | 368
Completed | 342
Not Completed | 26
Not completed — Technical Failure (No Test Device) | 26
Period: 36-Month Closure Evaluation
Arm/Group | Test Device
Started | 342
Completed | 278
Not Completed | 64
Not completed — Test Device Removal | 2
Not completed — Missed Echocardiograph | 62

BASELINE CHARACTERISTICS:
Arm/Group | Test Device
Number analyzed (Participants) | 400
Age, Continuous [Median (Full Range); unit: years] | 6.9 [1.3 to 79.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234
  Male | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55
  Not Hispanic or Latino | 319
  Unknown or Not Reported | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 16
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 45
  White | 286
  More than one race | 6
  Unknown or Not Reported | 45
Region of Enrollment [Number; unit: participants]
  United States | 400
Height [Median (Full Range); unit: cm] | 122.0 [40.5 to 188.0]
Weight [Median (Full Range); unit: kg] | 25.0 [9.0 to 133.6]
Hypertension [Count of Participants; unit: Participants]
  Current | 18
  Previous/Never | 382
Diabetes Mellitus [Count of Participants; unit: Participants]
  Current | 13
  Previous/Never | 387
Cigarette Smoking [Count of Participants; unit: Participants]
  Current | 7
  Previous | 8
  Never | 385
Headaches [Count of Participants; unit: Participants]
  Current | 15
  Previous/Never | 385
Migraines [Count of Participants; unit: Participants]
  Current | 15
  Previous/Never | 385
Cardiac Arrhythmia History [Count of Participants; unit: Participants]
  Current | 13
  Previous/Never | 387
Stop Flow Balloon Defect Size [Median (Full Range); unit: mm] — Population: Enrolled subjects with non-missing measurement
  mm
    number analyzed (Participants) | 393
    (all) | 12.0 [4.5 to 17.5]
Multiple Fenestrations [Count of Participants; unit: Participants] | 94
Atrial Septal Aneurysm [Count of Participants; unit: Participants] | 31
Septal Length [Median (Full Range); unit: mm] — Population: Enrolled subjects with non-missing measurement
  mm
    number analyzed (Participants) | 396
    (all) | 34.0 [6.0 to 64.0]
Anterior-Superior Aortic Rim Length [Median (Full Range); unit: mm] — Population: Enrolled subjects with non-missing measurement
  mm
    number analyzed (Participants) | 396
    (all) | 5.0 [0.0 to 24.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With 6-Month Composite Clinical Success
Description: Among subjects with attempted study device closure, the number of subjects who satisfy all of the following components:
  1. Technical Success: Successful deployment and retention at conclusion of index procedure of a GORE® CARDIOFORM Septal Occluder
  2. Safety Success:
     * Freedom from any Serious Adverse Event (SAE) through 30 days post-procedure
     * Freedom from device events (post-procedure embolization, device removal, or other device reintervention) from completion of the implant procedure through 6 months (195 days) post-procedure
  3. Closure Success: A clinical residual defect status of occluded or clinically insignificant as determined by the Echo Core Lab at the 6-month evaluation
Time Frame: 6 months
Population: All enrolled subjects with 6-month clinical success evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 368
Participants | 332
Statistical Analysis 1: Comparison: Test Device; Test null hypothesis of inferiority of test device (test) compared to historical device (control). H0: Pc - Pt ≥ Δ vs H1: Pc - Pt < Δ, where Pt and Pc are true proportions of 6-month clinical success for test and control, respectively, and Δ is the non-inferiority margin. Given Nc = 253, then Nt = 135 test subjects provides 86% power to reject H0 with 95% confidence if Δ = 0.10 and Pc = Pt = 0.866 under H0; Test type: Non-Inferiority — Non-inferiority margin based on 1) the lower 95% confidence bound (= 0.82) for estimated 6-month composite Clinical Success for the historical device (219/253=0.866), and 2) a worst-case analysis of 6-month composite Clinical Success for the historical device (0.81, assuming the 18 subjects with missing echo evaluations were failures); p < 0.0001, 2-sample binomial proportions test — A priori 1-sided alpha = 0.05; Risk Difference (RD) = -0.0366, 95% CI 1-sided [upper limit 0.007] — Difference is control - test. Confidence interval is the upper one-sided 95% Wald confidence interval

2. Secondary Outcome: Number of Subjects With Technical Success
Description: Among subjects with attempted study device closure, the number of subjects with successful deployment and retention at conclusion of index procedure of a GORE® CARDIOFORM Septal Occluder
Time Frame: During procedure; median duration 68 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 400
Participants | 374

3. Secondary Outcome: Number of Subjects With Procedure Success
Description: Among subjects with attempted study device closure, the number of subjects with technical success and less than or equal to 2 mm residual shunt of the target ASD at conclusion of the index procedure.
Time Frame: During procedure; median duration 68 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 400
Participants | 364

4. Secondary Outcome: Number of Subjects With 30-day SAE
Description: Among subjects with attempted study device closure, the number of subjects experiencing one or more serious adverse events (SAEs) within 30 days post-index procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 400
Participants | 7

5. Secondary Outcome: Number of Subjects With 6-Month Closure Success
Description: Among subjects with technical success, the number of subjects with clinical residual defect status of occluded or clinically insignificant as determined by the Echo Core Lab at the 6-month evaluation.
Time Frame: 6 months
Population: Enrolled subjects with technical success and 6-month clinical residual defect status evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 342
Participants | 338

6. Secondary Outcome: Number of Subjects With 12-Month Closure Success
Description: Among subjects with technical success, the number of subjects with clinical residual defect status of occluded or clinically insignificant as determined by the Echo Core Lab at the 12-month evaluation.
Time Frame: 12 months
Population: Enrolled subjects with technical success and 12-month clinical residual defect status evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 340
Participants | 337

7. Secondary Outcome: Number of Subjects With 36-Month Closure Success
Description: Among subjects with technical success, the number of subjects with clinical residual defect status of occluded or clinically insignificant as determined by the Echo Core Lab at the 36-month evaluation.
Time Frame: 36 months
Population: Enrolled subjects with technical success and 36-month clinical residual defect status evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Test Device
Number analyzed (Participants) | 278
Participants | 277

ADVERSE EVENTS:
Time Frame: 3 years (1,155 days: 1,095 days + 60-day window)
Description: SAEs follow definition of SAE from ISO 14155.
Arm/Group | Test Device
All-Cause Mortality (participants affected / at risk) | 0/400
Serious Adverse Events (participants affected / at risk) | 28/400
Other Adverse Events (participants affected / at risk) | 260/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Device (N=400)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Frenulum breve (Congenital, familial and genetic disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Medical device site thrombosis (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (3)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Croup infectious (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (2)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Penile adhesion (Reproductive system and breast disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Caesarean section (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Device (N=400)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 3 (3)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4)
Cardiac septal hypertrophy (Cardiac disorders) | 1 (1)
Dilatation atrial (Cardiac disorders) | 2 (2)
Extrasystoles (Cardiac disorders) | 2 (2)
Left ventricular dilatation (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 5 (5)
Nodal rhythm (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 16 (17)
Pericardial effusion (Cardiac disorders) | 3 (3)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 1 (1)
Pulmonary valve stenosis (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4)
Tricuspid valve incompetence (Cardiac disorders) | 3 (3)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Williams syndrome (Congenital, familial and genetic disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 2 (2)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Thyroid disorder (Endocrine disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Orbital cyst (Eye disorders) | 1 (1)
Strabismus (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Vitreous floaters (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9)
Dental caries (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (12)
Tongue disorder (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 24 (26)
Adverse drug reaction (General disorders) | 4 (4)
Asthenia (General disorders) | 2 (2)
Axillary pain (General disorders) | 1 (1)
Cardiac complication associated with device (General disorders) | 1 (1)
Chest discomfort (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Decreased activity (General disorders) | 1 (1)
Exercise tolerance decreased (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Generalised oedema (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Nodule (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 31 (38)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 18 (18)
Swelling (General disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Multiple allergies (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1)
Acute sinusitis (Infections and infestations) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 1 (2)
Bronchitis (Infections and infestations) | 5 (5)
Candida infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4)
Conjunctivitis (Infections and infestations) | 3 (3)
Croup infectious (Infections and infestations) | 5 (6)
Cystitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 6 (6)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 2 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2)
Impetigo (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 3 (3)
Lyme disease (Infections and infestations) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral viral infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 14 (14)
Otitis media acute (Infections and infestations) | 6 (7)
Otitis media chronic (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 8 (9)
Pharyngitis streptococcal (Infections and infestations) | 7 (7)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (3)
Rhinovirus infection (Infections and infestations) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 24 (27)
Urethritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 6 (7)
Viral rash (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 7 (7)
Vulvovaginitis (Infections and infestations) | 2 (2)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1)
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 1 (1)
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 5 (6)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 5 (5)
Incision site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 12 (12)
Incision site pain (Injury, poisoning and procedural complications) | 12 (12)
Incision site rash (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 3 (3)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 5 (6)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 4 (5)
Splinter (Injury, poisoning and procedural complications) | 1 (1)
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
Chest X-ray abnormal (Investigations) | 1 (1)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Infrapatellar fat pad inflammation (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Allodynia (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Dizziness postural (Nervous system disorders) | 5 (5)
Dysaesthesia (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 41 (45)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 10 (12)
Migraine with aura (Nervous system disorders) | 2 (2)
Migraine without aura (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (1)
Device issue (Product Issues) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Penile curvature (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (17)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3)
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Knee operation (Surgical and medical procedures) | 1 (1)
Air embolism (Vascular disorders) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1)
Carotidynia (Vascular disorders) | 1 (1)
Labile hypertension (Vascular disorders) | 1 (1)
Vascular dissection (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT01711983/Prot_SAP_000.pdf